CLINICAL TRIAL: NCT06520241
Title: The Effect of Stress, Anxiety, and Depression Experienced by Pregnant Women on Sleep Bruxism and Oral Health: Cross-sectional Study
Brief Title: The Effect of Stress, Anxiety, and Depression Experienced by Pregnant Women on Sleep Bruxism and Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Assist. Prof, Trakya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-SBB-0546
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Sleep Bruxism, Adult; Stress; Depression; Anxiety; Pregnancy Related; Oral Disease
MeSH Terms: conditions — Sleep Bruxism; Depression; Anxiety Disorders; Mouth Diseases | interventions — Gravidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pregnant — Data were collected using the Personal Information Form, Depression-Anxiety-Stress Scale (DASS-21), and Oral Health Impact Scale (OHIP-14-TR).

SUMMARY:
Background The oral health of pregnant women affects not only the systemic health of the mother but also the birth outcome of the fetus. Therefore, oral health management of pregnant women is important for both maternal and fetal health.

Objectives The study aimed to examine the effects of stress, anxiety, and depression experienced by pregnant women on sleep bruxism and oral health.

Methodology This cross-sectional study was conducted between September and November 2023 on 321 pregnant women who volunteered to participate in the study by posting on social media forum pages via the web. Data were collected using the Personal Information Form, Depression-Anxiety-Stress Scale (DASS-21), and Oral Health Impact Scale (OHIP-14-TR). Descriptive statistical methods, the Kruskal-Wallis test, Mann-Whitney-U test, and Spearman correlation test were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over the age of 18 who were pregnant, diagnosed with sleep bruxism, and who could read and write were included in the study.

Exclusion Criteria:

* Women who refused to participate in the study, who could not be contacted, who had serious dental health problems in the last six months, who had dentures, who had serious stress disorder in the last six months, who filled out the data collection form incompletely, who had hearing-vision problems or intellectual disability, and who had diagnosed psychological illness were not included in this study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 321 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Depression-Anxiety-Stress Scale | 1 day (collected once)
  Sarıçam (2018) adapted the scale developed by Lovibond and Lovibond (1995) into Turkish. In the scale consisting of depression, anxiety, and stress sub-dimensions, each sub-dimension consists of seven items. Scale items are scored from 0 to 3 (0=never and 3=always). Scores between 0 and 21 can be obtained from the scale sub-factors. Higher scores indicate higher levels of depression, anxiety, and stress.
Oral Health Impact Scale | 1 day (collected once)
  Oral Health Impact Scale (OHIP-14) with an internal consistency coefficient (Cronbach alpha) of 0.74, which was conducted by Başol et al. in 2014 for Turkish validity and reliability. The scale consists of 14 items with a 5-point Likert response scale (never-0; rarely-1; sometimes-2; often-3; very often-4) and seven subscales, each consisting of two items: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The total score obtained from the scale is obtained by summing the scores given to each item, and the total scale score range varies between 0 and 56.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided